CLINICAL TRIAL: NCT05941221
Title: Effect of Pericapsular Nerve Group (PENG) Block for Perioperative Analgesia in Geriatric Patients With Hip Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lydia edward aziz zakhary, Principal Investigator, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: pericapsular nerve group block
Record Dates: First submitted 2023-06-24; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Dental Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental): patients will receive pericapsular nerve group (PENG )block through ultrasound at the end of the surgery.
  Interventions: Procedure: pericapsular nerve group (PENG) block

INTERVENTIONS:
Procedure: pericapsular nerve group (PENG) block — patients will receive PENG block through ultrasound. The regional block was performed with the patient in the supine position. A curvilinear low-frequency ultrasound probe (2-5MHz) was initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed . A 22-gauge, 80-mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution was injected in 5-mL increments while observing for adequate fluid spread in this plane for a total volume of 20 mL bupivacaine 0.25%.

SUMMARY:
the goal of this clinical trial is to evaluate the analgesic effect of pericapsular nerve group (PENG) block in elderly patients with hip fractures undergoing hip surgery .

and to evaluate its effect in reducing post operative complications .

DETAILED DESCRIPTION:
all patients meeting the inclusion criteria will be informed about the study goal , methods and procedure in clear language. a written informed consent will be taken.

All patients ,once arrived to the OR, monitor will be attached, spinal anesthesia will be performed as follows, after sterilization of the back with bovidon iodine, local anesthesia 3cc of lidocaine 20% will be injected at the level of L3-L4 spine , then injection of 17 mg bupivacaine 0.5% through a 25 spinal needle.

At the end of surgery,all patients will receive PENG block through ultrasound. The regional block was performed with the patient in the supine position. A curvilinear low-frequency ultrasound probe (2-5MHz) was initially placed in a transverse plane over the AIIS and then aligned with the pubic ramus by rotating the probe counterclockwise approximately 45 degrees. In this view, the IPE, the iliopsoas muscle and tendon, the femoral artery, and pectineus muscle were observed. A 22-gauge, 80-mm needle was inserted from lateral to medial in an in-plane approach to place the tip in the musculofascial plane between the psoas tendon anteriorly and the pubic ramus posteriorly. Following negative aspiration, the local anesthetic solution was injected in 5-mL increments while observing for adequate fluid spread in this plane for a total volume of 20 mL bupivacaine 0.25%.

ELIGIBILITY:
Inclusion Criteria:

* patients must age 60 years or more .
* patients must belong to american society of anesthesiologists (ASA) classification class II or III

Exclusion Criteria:

* age < 60 years
* ASA IIII
* refusal of peripheral nerve block
* infection at the site of injection
* coagulopathy INR > 1.8
* platelets count < 50,000
* known allergy to used medications.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
post operative analgesic effect of PENG block | 24 hours
  evaluate the analgesic effect of PENG block in the post operative period both at rest and with movement using the Visual analog scale for pain

SECONDARY OUTCOMES:
post operative complications | 24 hours
  evaluate the effect of PENG block in reducing post operative complications like incidence of delirium using RAMSAY score

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Lin DY, Brown B, Morrison C, Fraser NS, Chooi CSL, Cehic MG, McLeod DH, Henningsen MD, Sladojevic N, Kroon HM, Jaarsma RL. The Pericapsular Nerve Group (PENG) block combined with Local Infiltration Analgesia (LIA) compared to placebo and LIA in hip arthroplasty surgery: a multi-center double-blinded randomized-controlled trial. BMC Anesthesiol. 2022 Aug 6;22(1):252. doi: 10.1186/s12871-022-01787-2. PMID 35933328
- [Background] Ying H, Chen L, Yin D, Ye Y, Chen J. Efficacy of pericapsular nerve group block vs. fascia iliaca compartment block for Hip surgeries: A systematic review and meta-analysis. Front Surg. 2023 Feb 10;10:1054403. doi: 10.3389/fsurg.2023.1054403. eCollection 2023. PMID 36843984